CLINICAL TRIAL: NCT04730700
Title: Evaluation of Multi-Tined Expandable Electrode (MEE) Efficacy and Safety in Treatment of Lumbar Facet Arthropathy by Radiofrequency Neurotomies Compared to Conservative Medical Management.
Acronym: MEE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dawood Sayed, MD, Study Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00146448
Record Dates: First submitted 2020-12-22; First posted 2021-01-29 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Radiofrequency ablation (RFA) with MEE (Active Comparator): Radiofrequency ablation involves a minimally invasive procedural technique. It uses radiofrequency waves to burn the nerve causing pain. This nerve will no longer be able to send pain signals to your brain. For this study, the multi-tined expandable electrode needle will be used. This needle will result in a larger treatment area. This may result in better pain relief and longer lasting pain relief. If you undergo the radiofrequency ablation procedure you will have pain medication injected where the ablation will be done. The procedure will take about 20 mins to complete. You will be allowed to go home afterward.
  Interventions: Procedure: Radiofrequency Ablation with MEE
- Conventional Medical Management (CMM) Treatment Only (Active Comparator): Your current standard of care treatment may already consist of some CMM therapies. Standard of care includes a variety of intervention types such as medication, physical therapy, home exercise programs, back brace, walking aid, and chiropractic care.
  Interventions: Behavioral: Conventional Medical Management

INTERVENTIONS:
Procedure: Radiofrequency Ablation with MEE — RFA will be performed in the usual fashion utilizing the MEE instead of the RFA needles routinely used at each institution.
  Arms: Radiofrequency ablation (RFA) with MEE
Behavioral: Conventional Medical Management — Conventional medical management (CMM), which may include physical therapy, home exercise programs, pain medication, and other conservative therapies such as back brace, walking aid, and chiropractic care.
  Arms: Conventional Medical Management (CMM) Treatment Only

SUMMARY:
The purpose of this study is to better understand how people feel after a radiofrequency ablation standard of care surgery using a different type of needle (multi-tined expandable electrode/MEE) in comparison to receiving conventional medical management (CMM) techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Patients with pain lasting at least 6 months.
* Patients with history of non-radiating low back pain.
* Patient who had two diagnostic medial branch blocks (MBB) with significant (>50%) improvement on both injections.
* Patient has signed study-specific informed consent.
* Patient has the necessary mental capacity to participate and is physically able to comply with study protocol requirements.

Exclusion Criteria:

* Patient with low back pain with radiation or involvement of pain going into their legs below their knees.
* Patient did not receive satisfactory relief from diagnostic MBB (<50% relief).
* Patient is unable to receive radiation exposure.
* Patient is currently pregnant.
* Patient has a current local overlying low back or systemic infection.
* Patient currently receiving or seeking workers compensation, disability remuneration, and/or involved in injury litigation.
* Known or suspected drug or alcohol abuse.
* Diagnosed psychiatric disease (e.g., schizophrenia, major depression, personality disorders) that could interfere with study participation.
* Patient is participating in an investigational study or has been involved in an investigational study within 3 months prior to evaluation for participation.
* Patient has an implanted intrathecal pump or spinal neuromodulation device.
* Patient currently on daily oral morphine equivalent (OME) of 50.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The mean visual analog scale (VAS) between the two group | 12 months
  will be compared using an independent samples t-test

SECONDARY OUTCOMES:
Observe the incidence of complications associated with MEE while utilizing this device | 12 months
  Number of complications will be analyzed using Independent samples T-Test if there is a normal distribution of complications. In the event of a binary outcome for complications, Chi-square Test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Sayed, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States